CLINICAL TRIAL: NCT06281600
Title: A Double-blind, Crossover Intervention Study Using Human Milk Oligosaccharides (HMOs) to Improve Irritable Bowel Syndrome (IBS) Symptoms Through Targeting of the Gut Microbiota
Brief Title: An Intervention Study Using HMOs to Improve IBS Symptoms
Acronym: GUT-HEAL-IBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glenn Gibson (Other)
Collaborators: Royal Berkshire NHS Foundation Trust (Other Government)
Responsible Party: Sponsor-Investigator, Glenn Gibson, Professor of Food Microbiology, University of Reading
Organization: University of Reading (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC: 23/SW/0042; 326109 (Other: IRAS ID)
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Gut microbiome; IBS; Human milk oligosaccharides
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: This is a 16-week, randomised, placebo-controlled, double-blinded crossover trial. We aim to recruit 44 participants with IBS. These participants will be screened and classified into a particular IBS subtype. After a 14-day baseline period, participants will be randomised to orally consume either 5g of HMO for 28 days, or a placebo for 28 days. This will be administered at the University of Reading. All participants will then stop taking the product for 28 days (wash out period) and then swap treatment type and have 28 days of either placebo or HMO. This is then followed by another 14 days without any product. During the study, participants will be asked to complete a 24-hour food recall weeks 0 and 16. Additionally, participants will complete validated questionnaires (IBS-Symptom Severity Score, anxiety and depression score and Pittsburgh Sleep Quality Index (PSQI) every time they provide urine and faecal samples at each visit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Every individual involved in undertaking this trial will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo control arm (Placebo Comparator): Maltodextrin will be given as a white powder placebo for 4 weeks.
  Interventions: Dietary Supplement: Maltodextrin placebo
- HMO intervention arm (Experimental): HMOs will be given as a white powder for 4 weeks.
  Interventions: Dietary Supplement: Human milk oligosaccharide

INTERVENTIONS:
Dietary Supplement: Human milk oligosaccharide — 5g daily dose of HMOs.
  Other Names: HMOs
  Arms: HMO intervention arm
Dietary Supplement: Maltodextrin placebo — 5g daily dose of maltodextrin.
  Other Names: Placebo
  Arms: Placebo control arm

SUMMARY:
There is now strong evidence implicating the human gut microbiota in many gastrointestinal diseases, including irritable bowel syndrome (IBS). Importantly, this enteric population is susceptible to dietary intervention and represents an exciting target for the prevention and treatment of gut mediated disorders. This study will investigate microbial components and activities associated with the gut microbiome, using a global systems biology approach to explore the capacity of a human milk carbohydrate intervention in modulating this microbial community to target IBS, with the primary objective of improving IBS symptoms.

IBS is a highly prevalent gastrointestinal (GI) disorder with significant negative impact on quality of life of patients and high healthcare costs. Although prognosis of IBS is benign, it is a disorder that poses a considerable burden on the individual sufferer and society. Patients typically present with chronic abdominal pain and an altered bowel habit, frequently accompanied by bloating and distension. Often, IBS will afflict sufferers for life, with flares of activity followed by periods of remission. Incidence commonly peaks in the third and fourth decades of life.

IBS is suggested to be a disorder of gut-brain interaction, and alterations of the microbiota-host interactions at the mucosal border may cause symptoms such as those previously mentioned. Therefore, microbiota-targeted interventions may benefit some people with IBS by beneficially modulating the gut microbiome. Several studies have confirmed that prebiotics, such as galactooligosaccharides (GOS), are able to successfully stimulate gut bifidobacteria and alleviate symptoms in IBS. Prebiotics are defined as "a substrate that is selectively utilised by host microorganisms conferring a health benefit" [8]. These studies suggest that prebiotics may have potential as therapeutic agents in IBS.

Breastmilk is known to play a crucial role in the development of infants, providing key nutrients and immunological compounds important for initial protection against pathogens [9]. Among these compounds, human milk oligosaccharides (HMOs) represent the third most important component of breastmilk after lipids and lactose. HMOs have also been investigated for potential health benefits in adults, including their potential role as prebiotics for improved gut microbiota modulation.

Studies looking specifically at HMO interventions in humans with IBS are sparse. These include a phase II, parallel, RCT in 58 IBS volunteers by Iribarren et al. and an open-label trial with 245 IBS participants from 17 sites across USA by Palsson et al.. None have been sufficiently powered to a degree which could influence clinical practice, but crucially tolerability and safety profiles of HMOs investigated, to date, have been consistently high.

Using the global systems biology approach not yet applied to this research question, a pre-competitive approach to selecting a candidate HMO, and a crossover feasibility trial design, the investigators hope to forge a new direction in establishing the merits of HMO use in IBS.

This study will look specifically at patients with all IBS subtypes, an area where there is a real therapeutic gap and clinical need for safe, effective therapy to improve quality of life. Participants will be randomly allocated to be given either the HMO or a placebo, with neither the patient nor the researchers knowing which they are receiving (randomised and double blind design). They will take this HMO or placebo for 28 days (randomly distributed), and then stop taking it in a 'washout' period of 28 days, allowing the gut microbiota to return to baseline. Then, the participants will take the other intervention (placebo or prebiotic, whichever they did not take in the first half of the study) for 28 days, then have a further washout period of 14 days. The study will then be over.

With this proposal, the aim is to explore how HMOs affect the gut microbiota and whether they can do so in a manner that positively influences patients with IBS. The investigators also hope to develop molecular profiling as part of a research toolkit for gut microbiome-based HMO supplement studies.

DETAILED DESCRIPTION:
The hypothesis of this study is that dietary supplementation with human milk oligosaccharides (HMO) will result in clinically significant improvement in IBS symptoms compared to placebo.

The null hypothesis is that HMO supplementation will have no different effect on disease activity compared to placebo. The alterative hypothesis is that HMO supplementation may worsen disease activity.

In this crossover design trial, patient reported outcome measures will be collected before, during and after both the intervention and placebo periods and compared.

With respect to secondary outcomes, this trial will also seek to identify if the HMO causes a reduction in anxiety and depression (measured and scored using validated questionnaire, PHQ-ADS), improvement in sleep quality (measured through Pittsburgh Sleep Quality Index, PSQI validated questionnaire), and changes in faecal microbiota (using 16S rRNA sequencing of key bacterial populations, e.g. bifidobacteria), changes in stool bacterial metabolites (measured as change in stool SCFA levels).

This is a 16-week, randomised, placebo-controlled, double-blinded crossover trial. The investigators aim to recruit 44 participants with IBS. These participants will be screened and classified into a particular IBS subtype. After a 14-day baseline period, participants will be randomised to orally consume either 5g of HMO for 28 days, or a placebo for 28 days. This will be administered at the University of Reading. All participants will then stop taking the product for 28 days (wash out period) and then swap treatment type and have 28 days of either placebo or HMO. This is then followed by another 14 days without any product. During the study, participants will be asked to complete a 24-hour food recall weeks 0 and 16. Additionally, participants will complete validated questionnaires (IBS-Symptom Severity Score, anxiety and depression score and Pittsburgh Sleep Quality Index (PSQI) every time they provide urine and faecal samples at each visit. All samples will be analysed at the University of Reading with the exception of 16S rRNA sequencing (patient data anonymised) which will be carried out by collaborators in Switzerland.

Collection and data analysis of questionnaire data will be carried out at The University of Reading.

1H-NMR spectroscopy-based metabolic profiling studies: In this proposal, 1H-NMR spectroscopy will be applied to characterise global metabolic signatures from biological samples collected throughout the human trials, using standard one-dimensional NMR experiments. Gut microbiology and metabonomic data will be integrated using data fusion techniques (for example, bidirectional partial least squares multi-block data analysis) to generate mechanistic understanding of system-level changes and optimise extraction of clinically relevant molecular information. It is anticipated that this analysis will provide a measure of how prebiotic based intervention during the clinical trial has affected the human metabonome in a manner closer to 'health.' Data collected will be bacterial community profiles, volunteer questionnaires, NMR-based metabonomic data, microbial end products and patient symptoms. These data will mostly be numerical and in the form of Excel spreadsheets, but will also include spectra data files, raw sequence files and food diary records (MS word/REDCap). Software for data analysis will be SAS (Statistical Analysis Software). Only the metabonomic NMR spectroscopy and microbial sequencing data files will generate moderately large data volumes. The investigators will identify community standards for data formatting for eventual deposit in data repositories.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form.
* Adults (aged from 18 to 60).
* Diagnosis of irritable bowel syndrome by a clinician (according to the Rome IV criteria).
* Absence of gut conditions other than IBS.

Exclusion Criteria:

* Intake of an experimental drug within four weeks prior to study.
* Former participation in prebiotic, probiotic or laxative trials within the previous four weeks.
* Former participation in a dietary intervention within the previous four weeks.
* Use of antibiotics within the previous four weeks.
* Intake of other specific prebiotics (such as oligosaccharides e.g. inulin), or probiotics (e.g. live yoghurts, other fermented products), drugs active on gastrointestinal motility, or a laxative of any class, for four weeks prior to study.
* Women who are lactating, pregnant or planning pregnancy during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
IBS-SSS | Clinically significant improvement in patient symptoms as defined by a decrease in IBS-symptom severity scoring over 16-week trial duration.
  Irritable Bowel Syndrome Symptom Severity Score validated questionnaire. Each measure is rated from 0 to 100, with total scores ranging from 0 to 500.

SECONDARY OUTCOMES:
Change in anxiety and depression scores (ADS) | Over 16-week trial duration.
  Measured and scored using validated questionnaire, PHQ-ADS. The PHQ-ADS is the sum of the PHQ-9 and GAD-7 scores and thus can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology.
Improvement of the Pittsburgh Sleep Quality Index (PSQI). | Over 16-week trial duration.
  A validated questionnaire measuring sleep quality. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Changes in faecal microbiota e.g. Bifidobacterium | Over 16-week trial duration.
  16S rRNA sequencing of key bacterial populations.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Gibson, Prof., Study Director — The University of Reading
Locations (1):
- The University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanz Morales P, Wijeyesekera A, Robertson MD, Jackson PPJ, Gibson GR. The Potential Role of Human Milk Oligosaccharides in Irritable Bowel Syndrome. Microorganisms. 2022 Nov 25;10(12):2338. doi: 10.3390/microorganisms10122338. PMID 36557589